CLINICAL TRIAL: NCT04620408
Title: Study on the Food Effects of Oral SHR4640 Tablets in Healthy Volunteers (Single Center, Randomized, Open, Double Crossover)
Brief Title: Study on the Food Effects of Oral SHR4640 Tablets in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: SHR4640-110
Record Dates: First submitted 2020-11-03; First posted 2020-11-09 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — ruzinurad

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): The subjects in group A did not have breakfast at D1, then were given an SHR4640 tablet. The subjects in group A had a high-fat breakfast on D8. After eating 30min, the subjects in group A were given SHR4640 tablet.
  Interventions: Drug: SHR4640
- Group B (Experimental): Group B had high-fat breakfast on D1, no breakfast on D8, and the rest was the same as group A.
  Interventions: Drug: SHR4640

INTERVENTIONS:
Drug: SHR4640 — Subjects were randomly divided into the group A, B. On D1, D8, two groups of subjects were respectively given SHR4640 tablet.

SUMMARY:
The primary objective of the study is to evaluate the effect of food on the pharmacokinetics of SHR4640 tablets in healthy volunteers. The secondary objective of the study is to observe the safety of SHR4640 tablets in healthy subjects.

DETAILED DESCRIPTION:
Subjects were randomly divided into the group A, B. On D1, D8, two groups of subjects were respectively given SHR4640 tablet.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form before the start of the activities related to this trial, and be able to understand the procedures and methods of this trial, and be willing to strictly abide by the clinical trial plan to complete this trial.
2. Aged between 18 and 45 years old (including both ends, whichever is the time of signing the informed consent form), male.
3. Body weight ≥ 50 kg, and body mass index (BMI): 19-26 kg/m2 (both ends included).

Exclusion Criteria:

1. Have a fertility plan within 3 months after screening to the last medication, or refuse to use medically approved contraceptive methods.
2. Drug abusers or drug urine screening positive.
3. Smokers (average daily smoking 5 or more).
4. Those who consumed more than 25 grams of alcohol per day during the first month were screened or were positive for alcohol breath test.
5. Anyone who had eaten grapefruit or fruit juice products within 2 days before administration, any food or drink containing caffeine (such as coffee, tea, chocolate, cola or other caffeinated carbonated drinks, etc.) and foods or drinks rich in purine food or alcohol.
6. The researchers judged that the subjects had medical conditions that affected the absorption, distribution, metabolism and excretion of drugs or reduced compliance.
7. Those with sUA > 420 µmol / L during the screening period, or those with a previous history of hyperuricemia and / or gout.
8. Those with estimated glomerular filtration rate (eGFR) < 90 (mL/min/1.73 m²) during the screening period.
9. Those with urolithiasis indicated or suspected by B ultrasound during the screening period.
10. Those who were positive for hepatitis B surface antigen (HBsAg), anti-hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody or syphilis antibody within one month or during the screening period.
11. Any clinical history of serious illness or disease or condition that the researchers believe may affect the results of the trial, including, but not limited to, a history of circulatory, endocrine, nervous, digestive, urinary or hematological, immune, mental and metabolic diseases.
12. People with allergies, including those who are explicitly allergic to research drugs or any ingredient in research drugs, are allergic to any food ingredient or have special requirements for diet, and are unable to follow a uniform diet.
13. Screening those who have undergone any operation within the first 3 months, or who have not recovered after the operation, or who may have a plan for operation or hospitalization during the trial.
14. Those who donated blood (or lost blood) within the first 3 months and donated blood (or lost blood) more than 400 mL, or received blood transfusion.
15. Screen people who have participated in clinical trials of any drug or medical device within the previous 3 months.
16. Take any prescription drug, over-the-counter medicine, Chinese herbal medicine or dietary supplement within 2 weeks before the screening period.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Cmax | Day1 to Day11
  Maximum observed concentration,
AUC0-t | Day1 to Day11
  Area under the curve from the time of dosing Dosing time to the last measurable (positive) concentration.
AUC0-inf | Day1 to Day11
  Area under the curve from time 0 to infinity

SECONDARY OUTCOMES:
sUA | Day1 to Day11
  concentration of serum urine acid

CONTACTS AND LOCATIONS:
Overall Officials: Beibei Liang, PhD, Principal Investigator — General Hospital of the Chinese people's Liberation Army

IPD SHARING:
Plan to Share IPD: No